CLINICAL TRIAL: NCT05089864
Title: Outcomes and Safety in Patients Treated With STAR and Deferred Stenting After Unsuccessful CTO PCI
Brief Title: STAR and Deferred Stenting Study
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Collaborators: Asahi-Intecc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-122
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Coronary Occlusion; Coronary Stenosis; Coronary Restenosis
Keywords: chronic total occlusion; sub-intimal plaque modification
MeSH Terms: conditions — Coronary Occlusion; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early stent placement (Other): Stent placement 5-7 weeks post-STAR procedure
  Interventions: Other: Stent Placement Timing - Early
- Later stent placement (Other): Stent placement 12-14 weeks post-STAR procedure
  Interventions: Other: Stent Placement Timing - Late

INTERVENTIONS:
Other: Stent Placement Timing - Early — Stent placement 5-7 weeks after STAR procedure
  Arms: Early stent placement
Other: Stent Placement Timing - Late — Stent placement 12-14 weeks after STAR procedure
  Arms: Later stent placement

SUMMARY:
STAR is a minimal-risk pragmatic clinical trial of patients admitted for a CTO-PCI procedure. The overall objective of the STAR Study is to address the current gaps in knowledge regarding use of STAR during CTO-PCI, as a prospective, multi-center study of 150 participants with randomization of timing of staged PCI. Five sites will be selected to participate in STAR from a national network of highly experienced CTO-PCI centers across the United States.

DETAILED DESCRIPTION:
To date, there have been no studies that prospectively and systemically evaluated the efficacy and safety of STAR with deferred stenting and described the frequency of its use in the hybrid approach. The aim of this study is to address these current gaps in knowledge, including the frequency of use of STAR by experienced operators, the safety of its use, optimal timing of staged stenting and health status change associated with this procedure. This prospective study will enroll 150 patients undergoing elective PCI of native CTO utilizing the STAR technique and will subsequently randomize patients in a 1:1 fashion to early (5-7 weeks) and later (12-14 weeks) timing of subsequent stenting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled for a PCI procedure for at least one chronic total occlusion with TIMI antegrade flow of zero.
2. Subject is ≥ 18 years of age at the time of consent
3. The operator attempted STAR technique defined as knuckle guidewire across or into the CTO segment during the CTO PCI and is planned for a staged procedure.
4. English speaking due to follow up.

Exclusion Criteria:

1. The CTO segment is in a graft.
2. Female subjects with a positive quantitative or qualitative pregnancy test, in accordance with hospital policy.
3. Unable to participate in telephone follow-up

   1. Too hard of hearing to do follow-up by telephone or deaf.
   2. Incarcerated prisoner.
   3. History of dementia.
   4. Subjects without a way for contact by telephone for follow-up.
4. Previously enrolled in STAR.
5. Patient not a candidate for baseline and final angiography (CKD with eGFR<30).
6. The knuckled guidewire did not cross into the CTO segment during STAR attempt.
7. A stent was placed into the STAR segment during the Index Procedure.
8. Refused participation in the study.
9. Patient enrolled in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Staged Procedure Success | 14 weeks
  success of the staged stenting procedure will be core lab adjudicated and defined as TIMI 3 flow, no major side branch loss, and residual stenosis <30%

SECONDARY OUTCOMES:
Vessel patency at time of staged stenting procedure | 14 weeks
  number of distal branches, and the antegrade TIMI flow through the vessel, assessed by core-lab analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werner GS, Martin-Yuste V, Hildick-Smith D, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, di Mario C, Hovasse T, Teruel L, Bufe A, Lauer B, Bogaerts K, Goicolea J, Spratt JC, Gershlick AH, Galassi AR, Louvard Y; EUROCTO trial investigators. A randomized multicentre trial to compare revascularization with optimal medical therapy for the treatment of chronic total coronary occlusions. Eur Heart J. 2018 Jul 7;39(26):2484-2493. doi: 10.1093/eurheartj/ehy220. PMID 29722796
- [Background] Sapontis J, Salisbury AC, Yeh RW, Cohen DJ, Hirai T, Lombardi W, McCabe JM, Karmpaliotis D, Moses J, Nicholson WJ, Pershad A, Wyman RM, Spaedy A, Cook S, Doshi P, Federici R, Thompson CR, Marso SP, Nugent K, Gosch K, Spertus JA, Grantham JA. Early Procedural and Health Status Outcomes After Chronic Total Occlusion Angioplasty: A Report From the OPEN-CTO Registry (Outcomes, Patient Health Status, and Efficiency in Chronic Total Occlusion Hybrid Procedures). JACC Cardiovasc Interv. 2017 Aug 14;10(15):1523-1534. doi: 10.1016/j.jcin.2017.05.065. PMID 28797429
- [Background] Brilakis ES, Grantham JA, Rinfret S, Wyman RM, Burke MN, Karmpaliotis D, Lembo N, Pershad A, Kandzari DE, Buller CE, DeMartini T, Lombardi WL, Thompson CA. A percutaneous treatment algorithm for crossing coronary chronic total occlusions. JACC Cardiovasc Interv. 2012 Apr;5(4):367-79. doi: 10.1016/j.jcin.2012.02.006. PMID 22516392
- [Background] Hirai T, Grantham JA, Sapontis J, Cohen DJ, Marso SP, Lombardi W, Karmpaliotis D, Moses J, Nicholson WJ, Pershad A, Wyman RM, Spaedy A, Cook S, Doshi P, Federici R, Nugent K, Gosch KL, Spertus JA, Salisbury AC; OPEN CTO Study Group. Impact of subintimal plaque modification procedures on health status after unsuccessful chronic total occlusion angioplasty. Catheter Cardiovasc Interv. 2018 May 1;91(6):1035-1042. doi: 10.1002/ccd.27380. Epub 2017 Oct 25. PMID 29068126
- [Background] Hirai T, Grantham JA, Gosch KL, Patterson C, Kirtane AJ, Lombardi W, Nicholson WJ, Moses J, Karmpaliotis D, Salisbury AC. Impact of Subintimal or Plaque Modification on Repeat Chronic Total Occlusion Angioplasty Following an Unsuccessful Attempt. JACC Cardiovasc Interv. 2020 Apr 27;13(8):1010-1012. doi: 10.1016/j.jcin.2020.01.214. No abstract available. PMID 32327084
- [Background] Galassi AR, Boukhris M, Tomasello SD, Marza F, Azzarelli S, Giubilato S, Khamis H. Long-term clinical and angiographic outcomes of the mini-STAR technique as a bailout strategy for percutaneous coronary intervention of chronic total occlusion. Can J Cardiol. 2014 Nov;30(11):1400-6. doi: 10.1016/j.cjca.2014.07.016. Epub 2014 Jul 22. PMID 25442438
- [Background] Goleski PJ, Nakamura K, Liebeskind E, Salisbury AC, Grantham JA, McCabe JM, Lombardi WL. Revascularization of coronary chronic total occlusions with subintimal tracking and reentry followed by deferred stenting: Experience from a high-volume referral center. Catheter Cardiovasc Interv. 2019 Feb 1;93(2):191-198. doi: 10.1002/ccd.27783. Epub 2018 Nov 9. PMID 30411863
- [Background] Xenogiannis I, Choi JW, Alaswad K, Khatri JJ, Doing AH, Dattilo P, Jaffer FA, Uretsky B, Krestyaninov O, Khelimskii D, Patel M, Mahmud E, Potluri S, Koutouzis M, Tsiafoutis I, Jaber W, Samady H, Jefferson BK, Patel T, Megaly MS, Hall AB, Vemmou E, Nikolakopoulos I, Rangan BV, Abdullah S, Garcia S, Banerjee S, Burke MN, Brilakis ES. Outcomes of subintimal plaque modification in chronic total occlusion percutaneous coronary intervention. Catheter Cardiovasc Interv. 2020 Nov;96(5):1029-1035. doi: 10.1002/ccd.28614. Epub 2019 Dec 4. PMID 31797507
- [Derived] Azzalini L, Kearney K, Salisbury AC, Stone N, Gosch KL, Jones PG, Spertus JA, Pershad A, Nicholson W, Lombardi W, Wyman RM, Davies R, Grantham JA, Hirai T; STAR Study Group. Early vs Late Staged PCI After Subintimal Tracking and Re-Entry for Chronic Total Occlusions: A Randomized Trial. J Am Coll Cardiol. 2026 Jan 27;87(3):286-293. doi: 10.1016/j.jacc.2025.09.1598. Epub 2025 Nov 26. PMID 41295935
- [Derived] Hirai T, Kearney K, Azzalini L, Salisbury AC, Stone N, Gosch KL, Pershad A, Nicholson W, Lombardi W, Wyman RM, Davies R, Grantham JA; STAR Study Group. Optimal timing of staged percutaneous coronary intervention after subintimal tracking and re-entry: Rationale and design of the subintimal tracking and re-entry with deferred stenting study. Catheter Cardiovasc Interv. 2024 Sep;104(3):444-450. doi: 10.1002/ccd.31161. Epub 2024 Jul 24. PMID 39044659